CLINICAL TRIAL: NCT05867407
Title: A Prospective Pragmatic Cluster-Randomized Care-as-Usual Controlled Study to Evaluate the Impact of an ECG-Based AI Algorithm to Detect Low Left Ventricular Ejection Fraction on Diagnosis Rates of LVEF ≤40% in the Outpatient Setting
Brief Title: A Multicenter Pragmatic Implementation Study of ECG-AI-Based Clinical Decision Support Software to Identify Low LVEF
Acronym: AIM ECG-AI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative decision following adoption of a new ECG-AI implementation workflow and slower-than-anticipated enrollment. No safety concerns; no outcome analyses were performed.
Sponsor: Anumana, Inc. (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DOC-244
Record Dates: First submitted 2023-05-01; First posted 2023-05-22 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Ventricular Ejection Fraction

STUDY DESIGN:
Intervention Model Description: Clinicians in primary care practice groups will be consented for enrollment into the study. Practice groups that decide to participate in the study will be randomized to have the software available or to provide care as usual without the software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Anumana Low EF AI-ECG Algorithm (Experimental): Anumana Low EF AI-ECG Algorithm
  Interventions: Device: Anumana Low EF AI-ECG Algorithm
- Care-as-Usual (Other): Care-as-Usual
  Interventions: Other: Care-as-Usual

INTERVENTIONS:
Device: Anumana Low EF AI-ECG Algorithm — Clinician will have access to the Anumana Low EF AI-ECG algorithm via a link in the patient's electronic health record which will display results applied to patients' ECGs, as well as supporting information. Using the results of the algorithm, combined with the clinician's knowledge of patient-specific risk factors, the clinician will determine whether further evaluation is warranted.
  Arms: Anumana Low EF AI-ECG Algorithm
Other: Care-as-Usual — Clinicians will not have access to the Anumana Low EF AI-ECG algorithm and will provide care-as-usual.
  Arms: Care-as-Usual

SUMMARY:
A prospective, cluster-randomized, care-as-usual controlled trial to evaluate the impact of an ECG-based artificial intelligence (ECG-AI) algorithm to detect low left ventricular ejection fraction (LVEF) on diagnosis rates of LVEF ≤ 40% in the outpatient setting.

The objective of this study is to evaluate the impacts of an ECG-AI algorithm to detect low LVEF and an associated Medical Device Data System when used during routine outpatient care. The study will be conducted in 2 phases: feasibility assessment phase and clinical impact phase.

DETAILED DESCRIPTION:
The study is a prospective, cluster randomized, care-as-usual controlled trial that will be conducted at 6 sites in the USA.

Primary care clinicians and general cardiologists will be invited and consented to participate in the study. For clinicians that accept, practice groups will be randomized to receive access to and education about the Low EF AI-ECG software and encompassing software or to provide care-as-usual in the control group. The study will be conducted in two phases: a feasibility pilot to evaluate integration and usability followed by observational period(s) to evaluate clinical outcomes.

Analyses of the primary and secondary endpoints will be conducted on data from patients that meet the inclusion and exclusion criteria. The expected duration of the study is 12 months, including a feasibility phase (estimated 6 weeks) followed by a 3-month initial observation period with rolling observation count monitoring until the target number of patient encounters is reached, followed by a 90-day follow up period.

At the completion of the feasibility period, we will evaluate quantitative and qualitative outcomes to inform the following observational period(s).

Primary endpoints and exploratory endpoints will be assessed the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years or older (including females who are pregnant, breastfeeding and/or lactating)
* Digital ECG captured or available within site for ECG-AI analysis at point-of-care

Exclusion Criteria:

* Known history of LVEF ≤ 40%
* Known history of systolic heart failure
* Known history of heart failure with reduced ejection fraction
* Opted out of electronic health record-based research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11610 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Diagnosis rates of low ejection fraction of less than or equal to 40 percent by echocardiography compared to care-as-usual | 90 days
  Diagnosis rates of low ejection fraction of less than or equal to 40 percent by echocardiography compared to care-as-usual

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Lopez-Jimenez, MD, MSc, MBA, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Duke Health, Durham, North Carolina
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Jimenez F, Alger HM, Attia ZI, Barry B, Chatterjee R, Dolor R, Friedman PA, Greene SJ, Greenwood J, Gundurao V, Hackett S, Jain P, Kinaszczuk A, Mehta K, O'Grady J, Pandey A, Pullins C, Puranik AR, Ranganathan MK, Rushlow D, Stampehl M, Subramanian V, Vassor K, Zhu X, Awasthi S. A multicenter pragmatic implementation study of AI-ECG-based clinical decision support software to identify low LVEF: Clinical trial design and methods. Am Heart J Plus. 2025 Mar 21;54:100528. doi: 10.1016/j.ahjo.2025.100528. eCollection 2025 Jun. PMID 40276542